CLINICAL TRIAL: NCT06990191
Title: A Hybrid 1 Effectiveness-Implementation Trial of Partner-Assisted Prolonged Exposure for PTSD
Acronym: COOPERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: University of Minnesota (Other); Center for Veterans Research and Education (Other); Arizona Veterans Research and Education Foundation (Unknown); Lowcountry Center for Veterans Research (Unknown); Veterans Medical Research Foundation (Other); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Atlanta VA Medical Center (U.S. Federal Agency); Tampa VA Healthcare System (Unknown); San Diego Veterans Healthcare System (U.S. Federal Agency); Charleston VA Healthcare System (Unknown); Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura A. Meis, Principal Investigator, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT9425-24-1-0499
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Trauma-focused therapies; Prolonged exposure; Veterans; Integrative Behavioral Couples Therapy; couples; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Exposure (PE) (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure (PE)
- Partnered Prolonged Exposure (PPE) (Experimental)
  Interventions: Behavioral: Partnered Prolonged Exposure (PPE)

INTERVENTIONS:
Behavioral: Partnered Prolonged Exposure (PPE) — The PPE condition adapts the PE protocol with strategies from Integrative Behavioral Couples Therapy (an evidence-based couple therapy. PPE involves twice-weekly 60-minute sessions, with some sessions completed by both the Veteran and their partner while others are with the Veteran only.
  Arms: Partnered Prolonged Exposure (PPE)
Behavioral: Prolonged Exposure (PE) — The PE condition will follow the standardized PE manual and involve weekly 90-minute sessions and a 30-minute check-in attended only by the Veteran and the therapist.
  Arms: Prolonged Exposure (PE)

SUMMARY:
PTSD occurs in up to 17% of post-9/11 US Service Members and is associated with long-term functional impairment, family problems, unemployment, and suicidality. Trauma-focused therapies (TFTs), such as Prolonged Exposure (PE), result in significant relief for many. Yet, TFTs are not equally effective for everyone. An important minority (~40%) will retain their PTSD diagnoses after treatment, and many discontinue treatment prematurely, especially post-9/11 Service Members. TFTs are also more effective in addressing symptoms than psychosocial functioning. More work is needed to improve the consistency and potency of TFTs. Partnering with significant others may provide a powerful method for helping individuals get more out of their PTSD treatment. Observational research shows that relationship factors can help patients initiate, stay in, and experience greater benefit from PTSD treatment. Veterans that were surveyed experienced greater treatment gains when they shared more about their treatment with loved ones and when loved ones accommodated less for PTSD symptoms. Despite the promise of partner-involved interventions, there is no couples approach to PTSD treatment that has demonstrated superior outcomes to individual-only treatment models (i.e., TFTs). To address this gap, the investigators have completed a series of partner-assisted PTSD treatment studies, leading up the current proposal (Partnered PE, PPE). The investigators found that treatment completion rates were better than routine clinical care, and the treatment led to large improvements in participants' functioning, PTSD symptoms, and romantic functioning. For this proposed study, the primary objective is to conduct a randomized controlled trial (Research Level 3; larger-scale clinical trial) to test the superiority of PPE to standard PE among post 9/11 Veterans. The investigator's primary hypothesis is that PPE will lead to greater improvements in psychosocial functioning than standard PE. Secondary and tertiary aims examine posttreatment clinical outcomes (PTSD, depression) and intimate partner outcomes (relationship functioning, distress, caregiver burden, and psychosocial functioning), as well as examine strategies for PPE implementation. In exploratory aims, the investigators will examine the stability of group differences, treatment completion rates, the role military sexual trauma history, and treatment mechanisms.

DETAILED DESCRIPTION:
Background: PTSD occurs in up to 17% of post-9/11 US Service Members and is associated with long-term functional impairment, family problems, unemployment, and suicidality. Trauma-focused therapies (TFTs), such as Prolonged Exposure (PE), result in significant relief for many. Yet, TFTs are not equally effective for everyone. An important minority (~40%) will retain their PTSD diagnoses after treatment, and many discontinue treatment prematurely, especially post-9/11 Service Members. TFTs are also more effective in addressing symptoms than psychosocial functioning. More work is needed to improve the consistency and potency of TFTs. Partnering with significant others may provide a powerful method for helping individuals get more out of their PTSD treatment. Observational research shows that relationship factors can help patients initiate, stay in, and experience greater benefit from PTSD treatment. Veterans that were surveyed experienced greater treatment gains when they shared more about their treatment with loved ones and when loved ones accommodated less for PTSD symptoms. Despite the promise of partner-involved interventions, there is no couples approach to PTSD treatment that has demonstrated superior outcomes to individual-only treatment models (i.e., TFTs). To address this gap, the investigators have completed a series of partner-assisted PTSD treatment studies, leading up the current proposal (Partnered PE, PPE). In PPE, intimate partners attend weekly treatment sessions. The study uses strategies from Integrative Behavioral Couples Therapy (ICBT), an efficacious, acceptance-based martial therapy intervention, to help couples support each other during treatment. PPE strives to increase the potency of PE through (1) teaching partners to act as effective PE coaches at home and (2) helping couples discuss trauma-related concerns together, providing an additional laboratory for exposure-based learning. Pilot findings support the feasibility and effectiveness of PPE. Treatment completion rates were better than routine clinical care, and the treatment led to large improvements in participants' functioning, PTSD symptoms, and romantic functioning.

Objectives: Our primary objective is to conduct a randomized controlled trial (Research Level 3; larger-scale clinical trial) to test the superiority of PPE to standard PE among post 9/11 Veterans.

Aims: Our primary hypothesis is that PPE will lead to greater improvements in psychosocial functioning than standard PE. Secondary and tertiary aims examine posttreatment clinical outcomes (PTSD, depression) and intimate partner outcomes (relationship functioning, distress, caregiver burden, and psychosocial functioning), as well as examine strategies for PPE implementation. In exploratory aims, the investigators will examine the stability of group differences, treatment completion rates, the role of military sexual trauma history, and treatment mechanisms.

Study Design: The study will use a mixed-method two-group Hybrid Type I effectiveness implementation RCT to determine the superiority of PPE to PE. The study team will run the study across three VAs (San Diego, Charleston, and Phoenix) over four-years. The Minneapolis VA will serve as a back-up site. 210 individuals with PTSD and their intimate partners will be randomized to PPE or PE and assessed at baseline, mid-treatment, posttreatment, 3-, and 6-mos posttreatment. The study team will conduct qualitative interviews with study participants, therapists, and clinical administrators to assess barriers and facilitators to PPE implementation to guide future implementation work.

Clinical Impact: The influence of a successful course of PTSD treatment on an individual's life is considerable. However, among current and former Service Members, the most effective treatments for PTSD yield smaller effects and fewer individuals finish them. PPE is well poised to improve the potency of trauma-focused treatment to ensure PE promotes recovery from PTSD for more Service Members. The study team will also explore differences for those with a history of military sexual trauma. Additionally, partnering with significant others during PE can answer long-standing calls for family-centered PTSD care and extend the benefits of PTSD treatment to families. Family involvement in PTSD care is highly desired by Service Members, a fertile avenue for improving the outcomes for patients with PTSD, and a national priority. Such research is critical to military service retention and to the health of the entire military. If PPE is more effective than PE, this proposal could feed the growth of symptom-focused psychotherapies that largely exclude loved ones into systems-based interventions designed to lift the whole person within the context of their important relationships.

ELIGIBILITY:
Inclusion Criteria:

* Post-9/11 Veteran Enrolled in VHA
* 1 > mo stable medication
* Committed relationship 6+ months
* DSM-5-R PTSD Diagnosis

Exclusion Criteria:

* Imminent suicidality/homicidally
* Mania, psychosis, or severe substance use disorder, past 3 mos
* Severe cognitive impairment
* Severe intimate partner violence in last 6 months
* Fear of or intimidation by partner
* Partner screens positive for PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (IPF) | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  The primary outcome is Veterans' global functioning at posttreatment assessment. The subdimensions of global functioning that matter most to Veterans with PTSD are their relationships with intimate partners, family relationships, work performance, friend relationships, parenting, educational performance, and self-care functioning (e.g., maintaining personal hygiene, exercising, household chores, healthy eating). Outcomes will be measured using the Inventory of Psychosocial Functioning (IPF).

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline, posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes. follow-up, 6 month follow-up
  Gold standard, structured-clinical interview that assesses PTSD symptom severity.
PTSD Checklist for DSM-5 (PCL-5) | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures PTSD symptom severity.
Patient Health Questionnaire - 9 (PHQ-9) | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures depression severity

OTHER OUTCOMES:
Couples satisfaction index | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures romantic relationship satisfaction
Perceived Stress Scale | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures perceived stress.
Short Zarit Burden Interview | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures caregiver burden.
WHO Disability Assessment Schedule (WHO-DAS 2.0) | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Self-report instrument that measures psychosocial functioning.
Inventory of Psychosocial Functioning (IPF) - Romantic functioning scale on partners | Baseline, mid-treatment (between session 5-6), posttreatment (immediately after treatment closes), and 3-months and 6-months after treatment closes.
  Subscale from a self-report instrument (the IPF) that measures relationship functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Meis, PhD, Principal Investigator — University of Minnesota, National Center for PTSD, Minneapolis VA Healthcare System; Leslie Morland, PhD, Principal Investigator — National Center for PTSD; San Diego VA Healthcare System
Locations (4):
- United States (4):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - San Diego VA Healthcare System, San Diego, California
  - Minneapolis VA Healthcare System, Minneapolis, Minnesota
  - Charleston VA Healthcare System, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
In accordance with 38 USC 7332, this type of information will be kept confidential and will not be disclosed in presentations, publications, or any other dissemination of the study results, or to anyone outside of the IRB-approved study team. Deidentified datasets will be made available following study completion. Participants will be notified of this during informed consent.
Time Frame: Deidentified datasets will be made available following study completion.

REFERENCES:
- [Background] Cusack K, Jonas DE, Forneris CA, Wines C, Sonis J, Middleton JC, Feltner C, Brownley KA, Olmsted KR, Greenblatt A, Weil A, Gaynes BN. Psychological treatments for adults with posttraumatic stress disorder: A systematic review and meta-analysis. Clin Psychol Rev. 2016 Feb;43:128-41. doi: 10.1016/j.cpr.2015.10.003. Epub 2015 Nov 2. PMID 26574151
- [Background] Steenkamp MM, Litz BT, Hoge CW, Marmar CR. Psychotherapy for Military-Related PTSD: A Review of Randomized Clinical Trials. JAMA. 2015 Aug 4;314(5):489-500. doi: 10.1001/jama.2015.8370. PMID 26241600
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Taft CT, Watkins LE, Stafford J, Street AE, Monson CM. Posttraumatic stress disorder and intimate relationship problems: a meta-analysis. J Consult Clin Psychol. 2011 Feb;79(1):22-33. doi: 10.1037/a0022196. PMID 21261431
- [Background] Jakupcak M, Cook J, Imel Z, Fontana A, Rosenheck R, McFall M. Posttraumatic stress disorder as a risk factor for suicidal ideation in Iraq and Afghanistan War veterans. J Trauma Stress. 2009 Aug;22(4):303-6. doi: 10.1002/jts.20423. PMID 19626682
- [Background] Kessler RC. Posttraumatic stress disorder: the burden to the individual and to society. J Clin Psychiatry. 2000;61 Suppl 5:4-12; discussion 13-4. PMID 10761674
- [Background] Richardson LK, Frueh BC, Acierno R. Prevalence estimates of combat-related post-traumatic stress disorder: critical review. Aust N Z J Psychiatry. 2010 Jan;44(1):4-19. doi: 10.3109/00048670903393597. PMID 20073563